CLINICAL TRIAL: NCT05438238
Title: Clinical Efficacy of Virtual Reality for Acute Pain and Anxiety Management During Egg Retrieval for in Vitro Fertility Treatment
Brief Title: Virtual Reality for Acute Pain and Anxiety During Egg Retrieval for in Vitro Fertility Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VR-OPU
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2022-06

CONDITIONS: Infertility; In Vitro Fertilization; IVF; ART
Keywords: virtual reality; infertility; transvaginal oocyte retrieval; IVF, in vitro fertilization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: This study is a comparison between the current standard practice of performing an egg retrieval with paracervical block (PCB) and virtual reality that is added to the above mentioned standard practice of TVOR + PCB. The aim of the study is to find out whether this newer technology has an advantage for the patient, in terms of anxiety and pain reduction, by aid of questionnaires
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- investigational group A (Experimental): during TVOR +PCB addition of Oncomfort, commercially available Virtual Reality headset, consisting of headphones with smartphone glasses - see oncomfort.com/en, CE approval conform IEC62366-1:2015, EN 62304:2006/Amd1:2015, EN 82304-1:2015, EN 82304-1:2016, ISO 13485:2016, EN ISO 14971:2019, EN 60601-1-2:2015
  Interventions: Device: Oncomfort
- reference group (No Intervention): standard of care TVOR + PCB

INTERVENTIONS:
Device: Oncomfort — Virtual Reality
  Arms: investigational group A

SUMMARY:
This study is a comparison between the current standard practice of performing a transvaginal oocyte retrieval (TVOR) with paracervical block (PCB) and a relatively recently developed technology of virtual reality that is added to the above mentioned standard practice of TVOR + PCB. The aim of the study is to find out whether this newer technology has an advantage for the patient, in terms of anxiety and pain reduction or satisfaction.

DETAILED DESCRIPTION:
People who wish to become pregnant sometimes have to resort to in vitro fertilisation (IVF) treatment. IVF treatment consists of the injection of hormones on one hand, and the creation and transfer of embryos on the other, with a view to pregnancy. The first part, the hormonal ovarian stimulation, leads to an egg retrieval through the maturation trigger 36h before. On the one hand, people may be very anxious about the unknown procedure, as they do not know what to expect. Due to the fertility problems and fertility treatments with its disappointments, there is also a psychological burden to be taken into consideration. On the other hand, people may experience this procedure as painful, although this varies greatly. Scientific studies show that 90% of women are comfortable during transvaginal oocyte retrieval under local anaesthetic and do not want additional painkillers.

Virtual reality has emerged in recent years as an alternative non-pharmacological treatment that has proven to be effective in treating burns, postpartum episiotomy suturing or in paediatric care.

The aim of this study is to investigate the alternative treatment (Virtual Reality glasses) for its effectiveness in treating anxiety and pain while undergoing transvaginal oocyte retrieval. The Virtual reality headmounted glasses by Oncomfort, CE certified,is a set of headphones with a smartphone screen that offers image and sound as a treatment, during the transvaginal oocyte retrieval, i.e. about 20-30 minutes.

Questionnaires will be filled out by the patients and the physician to evaluate expectations, fear and pain.

Prior to the TVOR, the patient will fill out the pre-operative questionnaire, which will interview their baseline fear, anxiety and expectations. Each patient is instructed on the use of the standard 100mm linear visual analog scale (VAS) with 0 as no pain and 10.0 as the worst pain imaginable.

In their room, after the TVOR, the patient will receive a second questionnaire (within 4h after oocyte retrieval, before leaving the hospital) about how the subject has experienced the exam, in general, at the worst moment, how attractive and immersive the VR was, and whether she would want to use the VR again.

Five days after the egg retrieval, the patient receives a third and last questionnaire on the experiences of the remaining day of the egg retrieval as well as the following days.

ELIGIBILITY:
Inclusion Criteria:

* female
* ≥18 and ≤ 40 years of age
* undergoing fertility treatments
* undergoing egg retrieval as part of in vitro fertilization treatment
* only first ≤ 3 IVF cycles.
* Bilateral ovarian follicular response (>3 and <30 follicles)

Exclusion Criteria:

1. Hearing impairments and blindness
2. Motion sickness
3. Any known anatomical characteristics that may make performing the office procedure impossible.
4. Patients undergoing a general anesthesia or conscious sedation
5. lack of informed consent
6. Chronic alcohol/drug abusers
7. Transabdominal approach for retrieval
8. Patients undergoing oocyte retrieval for fertility preservation before cancer or genotoxic treatment - oncofertility preservation
9. allergy to medications used

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Transvaginal oocyte retrieval requires controlled ovarian hyperstimulation of ovaries
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Difference in visual analog scale score for Pain | 1/ pre-procedure baseline 2/ immediately after the procedure and 3/ 5days after TVOR
  change in pain experience, assessed using visual analog scale (VAS). VAS is a 100mm linear visual analog scale with 0 as no pain and 10.0 as the worst pain imaginable.

SECONDARY OUTCOMES:
Difference in visual analog scale score for anxiety | 1/ pre-procedure baseline 2/ immediately after the procedure and 3/ 5days after TVOR
  change in anxiety experience, assessed using visual analog scale (VAS). VAS is a 100mm linear visual analog scale with 0 as no fear and 10.0 as the worst fear imaginable/ dying of fear

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Blockeel, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- UZ Brussel CRG, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No
all data will be anonymized before sharing with statistician